CLINICAL TRIAL: NCT05872126
Title: Video Assisted Thoracoscopic Surgery (VATS) - Surgical Pleurodesis vs Tube Drainage in Management of Malignant Pleural Effusion (MPE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kareem Ahmed Hosny, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AssiutMedicCTS
Record Dates: First submitted 2023-05-13; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Malignant Pleural Effusion; Thoracic Cancer
Keywords: Malignant pleural effusion; VATS; PleurX; Abrasion
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Intervention Model Description: Randomised Clinical Trial with 2 groups; Case group for VATS mechanical abrasion and Control group for tube drainage
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VATS surgical pleurodesis (Other): Patients in whom we use VATS-surgical pleurodesis for malignant pleural effusion.
  Interventions: Procedure: VATS-Surgical pleurodesis
- Tube drainage (Other): Patients in whom we use tube drainage for malignant pleural effusion.
  Interventions: Procedure: Tube Drainage

INTERVENTIONS:
Procedure: VATS-Surgical pleurodesis — VATS drainage and surgical abrasion.
  Arms: VATS surgical pleurodesis
Procedure: Tube Drainage — Tube drainage for malignant pleural effusion
  Arms: Tube drainage

SUMMARY:
Malignant Pleural Effusion (MPE) is considered to be a common presentation at malignant tumors representing 15% of all cancer cases. It carries a burden on our patients with dyspnea being the most common symptom in most of cases.

Management of symptomatic malignant pleural effusion remains to be a point of debate. Data available from literature shows conflicting results lacking high quality evidence which necsscitates further research work. Options differs to include chemical pleurodesis using medical or surgical talc poudrage or slurry. Surgical intervention with abrasion pleurodesis or pleurectomy using VATS approach has been used in many studies. Using indwelling pleural catheters (IPCs) has also proved comparable efficacy at many clinical trials. In this study we want to help answering this question so that we can add to the current knowledge aiming to offer the best care for those patients

ELIGIBILITY:
Inclusion Criteria:

* 1-patients with symptomatic malignant pleural effusion. 2- symptomatic patients with shortness of breath. 3-Lung can be fully expanded.

Exclusion Criteria:

1. Patients with non symptomatic malignant pleural effusion
2. Pleural symphysis with no potentiality for re-expansion
3. Patients managed surgically through open thoracotomy.
4. Pleural effusion due to causes other than malignancy
5. Loculated malignant effusion judged by chest ultrasound
6. Trapped lung due to malignant pleural effusion assessed by multislice CT chest.,
7. .Refusal to share the research project and not to sign the consent.

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Total hospital stay | 3 months postoperative
  duration of hospital stay in days
duration of airleak | 3 months postoperative
  duration in days

SECONDARY OUTCOMES:
Status of performance | 3 months
  patient reported outcome through a pre-prepared questionnaire
mortality | '3 months
  Rate of mortality
Failure of management | 3 months
  time to re-collection

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university heart hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided